CLINICAL TRIAL: NCT06944457
Title: A Phase I, Open-label, Single-center, Dose-escalation and Dose-finding Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of MPD-1 in Patients With Advanced Solid Tumor
Brief Title: Clinical Trial to Evaluate the Safety, Tolerability and Pharmacokinetics of MPD-1 in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pharosgen Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MPD-1_P1_01
Record Dates: First submitted 2024-11-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Cancer; Solid Tumor Cancer; Biomarkers
Keywords: PTEN Loss; KRAS mutation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: conventional 3+3 design with 4 arms (cohorts) to find RP2D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MPD-1 treatment (Experimental)
  Interventions: Drug: MPD-1

INTERVENTIONS:
Drug: MPD-1 — It is a prodrug that uses Doxorubicin to target KRAS mutant/ PTEN loss advanced cancer.

SUMMARY:
A Phase I, Open-label, Single-center, Dose-escalation and Dose-finding Clinical trial to evaluate the safety, tolerability and pharmacokinetics of MPD-1 in patients with advanced solid tumor

ELIGIBILITY:
Inclusion Criteria:

1. 19 to 75 years of age
2. A histologically or cytologically confirmed, metastatic or unresectable advanced solid tumor patient who has used all available existing standard therapy but tumor progression is confirmed and further treatment tool is absent, or patient showing resistant or inadequate to standard therapy.
3. KRAS mutation or PTEN loss is confirmed in tumor tissues prior to screening, and there is a documented record of this
4. Patients without the history of administration of anthracycline drugs and/or anthracene
5. Patients with at least one measurable or unmeasurable but assessable lesion in accordance with Response Evaluation Criteria in Solid Tumors Criteria (RECIST) 1.1
6. In screening and C1D1, subjects with appropriate hematologic, kidney, and liver function confirmed by the following laboratory test (one more laboratory test is permitted during the screening period)

<!-- -->

1. white blood cell (WBC) ≥ 3,500/mm3
2. absolute neutrophil count (ANC) ≥ 1,500/mm3 (without CSF administration within 2 weeks prior to C1D1)
3. platelets ≥ 100,000/mm3 (without transfusion within 2 weeks prior to C1D1)
4. hemoglobin (Hb) ≥ 10 g/dL (without transfusion within 2 weeks prior to C1D1)
5. total bilirubin ≤ 1.5 times the normal upper limit (However, in case of Gilbert syndrome, this patient can participate in this clinical trial regardless of the results of total bilirubin
6. aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 times the normal upper limit (five times of the normal upper limit in case of liver metastasis)
7. albumin ≥ 2.5 g/dL
8. serum creatinine ≤ 1.5 times the normal upper limit
9. INR ≤ 1.5 times the normal upper limit 7) Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 8) Patients with an expected survival period of more than 12 weeks 9) Patients who have recovered from previous therapy-related adverse event to Common Terminology Criterion for Adverse Events (CTCAE) version 5.0 grade 1 or below or to C1D1 levels (However, sHair loss (regardless of grade), subjects can be enrolled if they have with hair loss (regardless of grade) or peripheral neuropathy below grade 2 or laboratory test results show that they do not meet the exclusion criteria) can be enrolled.) 10) Patients, who after understanding all the relevant information of this clinical trial, decides to participate, and voluntarily signed a written agreement.

Exclusion Criteria:

1. Within 4 weeks prior to the C1D1, subjects who underwent surgery, chemotherapy (cytotoxic, targeted antitumor drugs), immunotherapy, biological or hormonal therapy, or radiation therapy at areas exceeding 30% of bone marrow for the treatment of this clinical trial's target disease
2. Participation in other interventional clinical trials (administration of investigational new drugs or use of investigational medical devices) within 4 weeks prior to C1D1
3. Subjects who are identified with the following comorbidities during screening

   - Clinically significant symptomatic or uncontrolled central nervous system metastasis (but can participate in this clinical trial if systemic corticosteroids have not been administered for more than 2 weeks prior to C1D1 and the condition is stable)
   * Heart disease that could affect this clinical trial (left ventricular ejection fraction (LVEF) <50%, congestive heart failure with New York Heart Association (NYHA) class II or higher, history of myocarditis, myocardial infarction or unstable angina within 24 weeks before C1D1, uncontrolled cardiac dysrhythmia by appropriate medication, coronary artery disease, etc.)
   * History of thrombosis (e.g., thrombophlebitis, etc.)
   * Uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg)
   * Clinically significant ascites
   * Subjects who are infected with or carrying hepatitis B virus (HBV) or hepatitis C virus (HCV)* * When screening, serology tests show that any one of the following is positive: hepatitis B surface antigen (HBsAg), hepatitis B core antibody-immunoglobulin M (HBcAb-IgM), and hepatitis C virus antibody (HCV Ab) (However, if the HCV Ab test result is suspected to be false positive or positive due to past infection, HCV RNA test may be performed at each institution under the judgement of investigator and the HCV Ab and RNA test results are integrated to decide whether HCV is infected.)
4. The following medical history is identified during screening

   * Chickenpox or varicella zoster infection within 12 weeks prior to C1D1
   * Uncontrolled active infectious diseases including known human immunodeficiency virus (HIV) positives
5. Subjects with a history of administration of the following drugs during screening or C1D1

   * Vaccination against yellow fever within 4 weeks prior to C1D1
   * Penitoin within 1 week prior to C1D1
   * G-CSF administration to correct absolute neutrophil count (ANC) levels within 2 weeks prior to C1D1

     -- Transfusion of packed red cells or platelets to correct platelets or hemoglobin levels within 2 weeks prior to C1D1
   * Trastuzumab within 28 weeks prior to C1D1
6. Pregnant women, nursing mothers, and fertile women with plan for pregnancy
7. Fertile women or men who do not agree to abstain from sex or perform effective contraception methods for at least 24 weeks after the end of administration* [* Effective Contraception]

   * Hormone contraception (oral contraceptives, subcutaneous implants, etc.)

     * Intrauterine device (IUD) or implantation of an intrauterine system (IUS) ③ Infertility procedures or surgeries (vasectomy, bilateral oviduct ligation/excision, hysterectomy, etc.)

       * Double contraception (concurrent use of contraceptive methods from ①~③ and condoms for men or women) ⑤ Absolute abstinence: Based on investigator's judgment, thorough abstinence from sex is approved if the subject's age, occupation, lifestyle, or sexual orientation guarantee contraception. However, periodic abstinence (menstrual cycle, mucus method, symptomatic body temperature method, etc.), resection, and withdrawal method (coitus interruptus) are not recognized as appropriate contraception methods.
8. Subjects who have a history of allergies to doxorubicin or the excipient of MPD-1 or is suspicious of allergy
9. Subjects in a state of prohibiting, limiting, or disrupting the assessments specified in the clinical trial (e.g., a history of alcohol or drug abuse within two years prior to C1D1)
10. Subjects considered as unsuitable for participation in the clinical trial by the investigator (e.g., if the patient's health is unsuitable or participation in this clinical trial is not the best treatment for the patient)

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) Determination | From first treatment to the end of treatment at 18 weeks
  Number of participants experiencing dose-limiting toxicities (DLTs) during the DLT observation period (3 weeks, 1 cycle) following administration of MPD-1, as defined by CTCAE v5.0 criteria.
  • Unit of Measure: Number of participants with DLTs
Incidence of Treatment-Related Adverse Events | From first treatment to the end of treatment at 18 weeks
  Number of participants experiencing treatment-related adverse events, as assessed by CTCAE v5.0.
  • Unit of Measure: Number of participants
Electrocardiogram (ECG) QT Interval Prolongation | From first treatment to the end of treatment at 18 weeks
  Number of participants with QT interval prolongation (QTc > 450 ms for males, > 470 ms for females) on 12-lead ECG.
  • Unit of Measure: ECG QT interval

SECONDARY OUTCOMES:
Pharmacokinetic Outcome Measures | From first treatment (Cycle 1, Day 1) to one week after the first treatment (Cycle 1, Day 8)
  Peak Plasma Concentration: Cmax
Pharmacokinetic Outcome Measures | From first treatment (Cycle 1, Day 1) to one week after the first treatment (Cycle 1, Day 8)
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetic Outcome Measures | From first treatment (Cycle 1, Day 1) to one week after the first treatment (Cycle 1, Day 8)
  Tmax (Time to Maximum Concentration)
Pharmacokinetic Outcome Measures | From first treatment (Cycle 1, Day 1) to one week after the first treatment (Cycle 1, Day 8)
  t1/2 (Elimination Half-Life)
Pharmacokinetic Outcome Measures | From first treatment (Cycle 1, Day 1) to one week after the first treatment (Cycle 1, Day 8)
  CL (Clearance)

CONTACTS AND LOCATIONS:
Overall Officials: Sangyoon Kim, MD, PhD, Study Director — Pharosgen Co.,Ltd
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided